CLINICAL TRIAL: NCT00003846
Title: Treatment of High Risk Central Nervous System Embryonal Tumors With Conventional Radiotherapy and Intensive Consolidation Chemotherapy With Peripheral Blood Progenitor Cell (PBSC) Support
Brief Title: Radiation Therapy, Chemotherapy, and Peripheral Stem Cell Transplantation in Treating Patients With Primitive Neuroectodermal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99702; COG-99702 (Other: Children's Oncology Group); CCG-99702 (Other: Children's Cancer Group); CDR0000067006 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cyclophosphamide; Thiotepa; Triethylenephosphoramide; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: thiotepa; Drug: vincristine sulfate; Procedure: bone marrow ablation with stem cell support; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: Neupogen®; G-CSF; NSC#614629
Drug: carboplatin
  Other Names: Paraplatin®; CBDCA; NSC#241240
Drug: cyclophosphamide
  Other Names: Cytoxan®; Neosar®; Procytox®; CPM
Drug: thiotepa
  Other Names: TRIETHYLENETHIOPHOSPHORAMIDE; THIOPLEX®; TEPA; NSC# 6396
Drug: vincristine sulfate
  Other Names: Oncovin®; Vincasar®; leucocristine; VCR; NSC# 67574
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of radiation therapy and chemotherapy and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy, chemotherapy and peripheral stem cell transplantation in treating patients with primitive neuroectodermal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of postradiotherapy high-dose consolidation chemotherapy with peripheral blood stem cell (PBSC) support in patients with high-risk primitive neuroectodermal tumors.
* Determine the safety of delaying radiotherapy by approximately one month in these patients.
* Determine the maximum tolerated dose of thiotepa in these patients.
* Determine the toxic effects of intensive chemotherapy with PBSC support in these patients.
* Assess the time to hematopoietic recovery after PBSC infusion when intensive chemotherapy is used after craniospinal radiotherapy in these patients.
* Determine the overall and event-free survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of thiotepa during consolidation therapy.

* Induction: Within 31 days of initial surgery, patients receive induction therapy comprising vincristine IV on day 0, cyclophosphamide IV over 2 hours on days 0 and 1, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 2 and continuing for at least 7-10 days. Peripheral blood stem cells (PBSC) are then collected.
* Chemoradiotherapy: After blood cell counts recover, and within 28 days of starting induction, patients begin chemoradiotherapy. Patients receive vincristine IV once weekly for 8 doses. Radiotherapy is administered 5 days a week, for 6 weeks, beginning within the same week as the start of vincristine.
* Consolidation: Therapy begins 4-6 weeks after the last radiation treatment in the absence of disease progression. The first and third course are the same and comprise vincristine IV on day 0, carboplatin IV over 1 hour on days 0 and 1, thiotepa IV over 3 hours on days 2-4, and G-CSF SC daily beginning on day 7. PBSC are reinfused on day 7. The second course comprises vincristine IV on day 0, carboplatin IV over 1 hour on days 0 and 1, cyclophosphamide IV over 2 hours on days 2 and 3, and G-CSF SC daily beginning on day 5. PBSC are reinfused on day 5. Each course lasts 21 days.

For consolidation therapy, cohorts of 6-12 patients each receive escalating doses of thiotepa until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 12 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 24-56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primitive neuroectodermal tumor (PNET) of one of the following types:

  * Atypical teratoid/rhabdoid tumor
  * Medulloblastoma
  * Desmoplastic medulloblastoma
  * Ependymoblastoma
  * Medullomyoblastoma
  * Spongioblastoma
  * Spongioblastoma polare
  * Primitive polar spongioblastoma
  * Medulloepithelioma
  * Neuroblastoma
  * Pineoblastoma
* Posterior fossa PNET must be M1-3 or M0 with greater than 1.5 cm2 residual disease
* Non posterior fossa PNET and other types must be M0-3

  * If M3, must show clear evidence of tumor on MRI
* No marrow involvement or other extraneural metastases
* No M4 disease
* No cord compression requiring emergency radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 150,000/mm^3 (no platelet transfusions)
* Hemoglobin at least 10 g/dL (red blood cell transfusions allowed)

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST or ALT less than 2.5 times ULN

Renal:

* Creatinine clearance or glomerular filtration rate at least 70 mL/min

Cardiovascular:

* Shortening fraction greater than 27% by echocardiogram OR
* Ejection fraction greater than 47% by MUGA

Pulmonary:

* FEV_1/FVC greater than 60% except for children who:

  * Are uncooperative
  * Have no dyspnea at rest
  * Have no exercise intolerance
  * Have pulse oximetry greater than 94% on room air

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Steroids for increased intracranial pressure allowed

Radiotherapy:

* See Disease Characteristics
* No prior urgent radiotherapy

Surgery:

* Not specified

Other:

* No prior therapy for tumor

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 1999-07; Primary Completion 2004-10 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: H. Stacy Nicholson, MD, MPH, Study Chair — OHSU Knight Cancer Institute
Locations (13):
- United States (13):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington